CLINICAL TRIAL: NCT03720574
Title: Efficacy and Safety of Lorcaserin and Behavioral Modification for Overweight and Obesity Management in Chinese Adult Obese Patients: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Lorcaserin and Behavioral Modification for Overweight and Obesity Management in Chinese Obese Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Reassess safety risks and benefits
Sponsor: Kanion & Huawe Medicine Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LWY17016C
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Obesity
Keywords: Overweight or Obesity Management; Behavioral Modification
MeSH Terms: conditions — Obesity; Overweight | interventions — lorcaserin; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lorcaserin 10 mg BID (Experimental): Lorcaserin 10 mg tablet each morning and evening
  Interventions: Drug: Lorcaserin 10 mg BID
- Matching Placebo BID (Placebo Comparator): Matching Placebo tablet each morning and evening
  Interventions: Drug: Matching Placebo BID

INTERVENTIONS:
Drug: Lorcaserin 10 mg BID — Lorcaserin 10 mg tablet each morning and evening for a duration of 48 weeks
  Arms: Lorcaserin 10 mg BID
Drug: Matching Placebo BID — Matching Placebo tablet each morning and evening for a duration of 48 weeks
  Arms: Matching Placebo BID

SUMMARY:
The purpose of this study is to assess the safety and weight loss effect of lorcaserin at the end of the first year of treatment (Week 48) in overweight and Chinese adult obese patients compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged from 18 to 65 years (inclusive).
* Able to walk and preform exercise program required by trial protocol.
* Body Mass Index (BMI) within the range of 30 to 45 kg/m2 (obese) with or without co-morbid conditions or greater than or equal to 27 and less than 30 kg/m2 (overweight) with at least one treated or untreated comorbid condition (hypertension, dyslipidemia, cardiovascular disease, untreated abnormal glucose metabolism, sleep apnea). For untreated co-morbid conditions, the condition must be considered by the Investigator as clinically stable.
* Prior to the study, patients should be able to voluntarily participate in this study and sign informed consent form approved by IRB/ICE

Exclusion Criteria:

* Not suitable to participate in the study in the opinion of the Investigator, including an existing physical or mental condition that prevents compliance with the protocol.
* Patients who had a history of Type 1 diabetes mellitus or confirmed diagnosis of Type 2 diabetes mellitus for more than 6 months.
* Recent history (within 1 years before entering the study) of major depression, anxiety, or other psychiatric disease requiring treatment with prescription medication (e.g., SSRI's, SNRI's [including buproprion], tricyclics, antipsychotics, lithium). Use of SSRI's and SNRI's (including buproprion) for reasons other than active psychiatric indications (e.g., migraine, weight loss, smoking cessation) must meet a 3-month washout.
* Total score on the Beck Depression Inventory-II (BDI-II) > 20.
* Binge Eating Scale score >17.
* History of epilepsy or other seizure disorder.
* Has done or anticipate Surgical procedure for the treatment of obesity (i.e., gastric bypass, gastric banding).
* Anticipation of surgery during the study period that may interfere with completion or compliance with the protocol.
* Uncontrolled hypertension after certain treatments, defined as systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥ 100 mmHg.
* History of valve replacement surgery or CABG or other invasive cardiovascular surgical procedure. A diagnostic cardiac catheterization does not exclude.
* History of Myocardial infarction(MI), Cerebral Vascular Accident(CVA), or transient ischemic attack(TIA). Reversible ischemic neurological deficits (RIND), cardiac arrhythmia requiring medical or surgical treatment within 3 months of screening.
* Major surgical procedure (intrathoracic, intracranial, intraperitoneal, liposuction) within 6 months of screening
* History of unstable angina
* History of congestive heart failure caused by insufficiency or stenosis of any heart valve
* History of pulmonary artery hypertension
* Symptomatic untreated congestive heart failure of any etiology (stably treated NYHA class I or II CHF of ischemic or hypertensive etiology is acceptable)
* History of organ/bone marrow transplantation
* Abnormal TSH lab value > 1.5x ULN
* Hyperthyroidism, including abnormal screening lab values with FT4 > ULN and TSH < LLN.
* Fasting triglycerides > 499 mg/dL(5.64 mmol/L) ,if elevated at Screening, but not on a subsequent re-check, patient will be eligible. Otherwise, patients can't be enrolled.
* LDL-cholesterol ≥ 190 mg/dL(4.92 mmol/L).
* HbA1c greater than 9.0%
* Fasting glucose > 270 mg/dL(11.0 mmol/L) ,if elevated at Screening, but not on a subsequent re-check, patient will be eligible. Otherwise, patients can't be enrolled.
* Clinically significant abnormal hepatic (e.g., AST or ALT > 2.5x ULN, or total bilirubin > 1.5x ULN) or renal function lab tests (e.g., creatinine > 1.25x ULN) suggestive of hepatic or renal impairment.
* Positive result of HIV, hepatitis B or hepatitis C screens.
* Malignancy within 5 years of the screening visit (except basal cell or squamous cell carcinoma with clean surgical margins).
* Treatment with over-the counter weight loss products or appetite suppressants (including herbal weight loss agents) within 1 month of the screening visit, or with a prescription anti-obesity drug (phentermine, sibutramine, orlistat) or lipid dissolving injections within 3 months.
* Over 3 days of treatment with oral or parenteral corticosteroids within 2 weeks of the screening visit.
* Recent history (within 2 years prior to the screening visit) of alcohol or drug abuse.
* Significant change in smoking habits within 3 months prior to screening.
* Participated in any clinical study with an investigational drug, biologic, or device within 3 month prior to screening.
* Significant change in diet or level of physical activity or change in weight of > 5 kg within 3 month prior to screening.
* Use of liquid weight loss diet within 6 months prior to screening.
* Disagree to continue to use an accepted method of birth control during and for at least 3 months after last study medication administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
5% responders | 48 weeks
  Proportion (%) of subjects who lose at least 5% of their baseline body weight at week 48

SECONDARY OUTCOMES:
Weight change | 48 weeks
  Change from baseline in body weight (kilograms) at week 48
10% responders | 48 weeks
  Proportion (%) of subjects who lose at least 10% of their baseline body weight at week 48
circumference and hip circumference change | 48 weeks
  Change from baseline in waist circumference and hip circumference (centimeters) at week 48
Blood Pressure change | 48 weeks
  Change from baseline in waist systolic/ diastolic blood pressure (mmHg) at week 48
Lipids change | 48 weeks
  Change from baseline in Lipids (total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides) (mmol/L) at week 48
CV Risk Markers change | 48 weeks
  Change from baseline in CV Risk Markers (CRP in μg/L, fibrinogen in g/L) at week 48
Glucose and HbA1c change | 48 weeks
  Change from baseline in fasting glucose (mmol/L) and HbA1c (%) at week 48
IWQOL-LITE score change | 48 weeks
  Change from baseline in IWQOL-LITE score at week 48

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Guo, Ph. D, Principal Investigator — Peking University First Hospital
Locations (9):
- China (9):
  - Bengbu Medical College First Affiliated Hospital, Bengbu, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Second Hospital of Changzhou, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Jinzhou Central Hospital, Jinzhou, Liaoning
  - Jinan Center Hospital, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No